CLINICAL TRIAL: NCT06183866
Title: Evaluation of the Exposure to Chemical Substances of Some of the Employees Working in a Household Waste Incineration Plant
Brief Title: Exposure to Chemical Substances Within Household Waste Incineration Plants
Acronym: Chem-Expo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8721
Record Dates: First submitted 2022-12-16; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2022-12

CONDITIONS: Exposure to Chemical Pollution, Occupational
Keywords: Chemical Pollution

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Employees of household waste incineration plants (UIOM) are exposed to multiple chemical substances that can pose a risk to their health.

The studies carried out find increases in certain toxic chemicals (heavy metals, dioxins), in the biological fluids of employees (blood, urine), in particular before the 2000s Another study conducted by Tait finds potential organic alterations.The investigators wish to complete the dissertation work with, in particular, an analysis of the quantitative elements of the exposure assessment (metrologies and biometrologies)

DETAILED DESCRIPTION:
The aim of the study is to evaluate the recorded chemical exposures of certain employees of a household waste incineration plant (UIOM) in order to deduce the risk to their health.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject currently working, or having worked in the Strasbourg waste incineration plant between 01/01/2013 and 01/09/2022 within the maintenance or operating team
* Subject not objecting, after being informed, to the reuse of their data for the purposes of this research
* Subject in whom one or more biometrologies (blood lead level measurement, urinary cadmium level measurement, urinary 1-hydroxypyrene level measurement) were performed

Exclusion criteria:

-Subject who expressed their opposition to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject currently working, or having worked in the Strasbourg waste incineration plant between 01/01/2013 and 01/09/2022 within the maintenance or operating team
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective evaluation of the identified chemical exposures of certain employees of a household waste incineration plant (UIOM) in order to deduce the risk to their health. | Files analysed retrospectively from 01 January 2013 to 01 September 2022 will be examined
  The study is based on a retrospective analysis of existing data in the files of patients treated by the occupational medicine department

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pathologie Professionnelle et Médecine du Travail - CHU de Strasbourg - France, Strasbourg, France